CLINICAL TRIAL: NCT00114335
Title: Prevalence of Impaired Renal Function in Medical Inpatients
Brief Title: Epidemiologic Data of Patients in a Teaching Hospital
Status: Completed | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Other Study IDs: LMWHplus_1
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Kidney Diseases; Obesity
Keywords: low molecular weight heparin; unfractionated heparin
MeSH Terms: conditions — Kidney Diseases; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This small cross-sectional epidemiological study is designed to evaluate the prevalence of the following parameters in hospitalized patients in a tertiary teaching hospital (medical department only):

* kidney insufficiency
* obesity
* use of unfractionated heparins / low molecular weight heparins
* other drugs effecting the hemostatic system

DETAILED DESCRIPTION:
This small cross-sectional epidemiological study is designed to evaluate the prevalence of the following parameters in hospitalized patients in a tertiary teaching hospital (medical department only):

* kidney insufficiency
* obesity
* use of unfractionated heparins / low molecular weight heparins
* other drugs effecting the hemostatic system

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized at the defined days (two days) at Kantonsspital Luzern, Department of Medicine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized at the defined days (two days) at Kantonsspital Luzern, Department of Medicine
Sampling Method: Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2005-05; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P Schmid, MD, Principal Investigator — Kantonsspital Luzern, Hematology; A G Fischer, MD, Study Director — Kantonsspital Luzern, Nephrology; W A Wuillemin, MD, PhD, Study Chair — Kantonsspital Luzern, Hematology
Locations (1):
- Kantonsspital Luzern, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Result] Schmid P, Fischer AG, Wuillemin WA. Prevalence of impaired renal function in medical inpatients. Swiss Med Wkly. 2007 Sep 8;137(35-36):514. doi: 10.4414/smw.2007.11903. No abstract available. PMID 17990139
- See also: Luzerner Kantonsspital, Hematology — http://www.ksl.ch/standorte/luzern/kliniken/medizin/haematologie.html
- See also: Luzerner Kantonsspital, Nephrology — http://www.ksl.ch/standorte/luzern/kliniken/medizin/nephrologie.html
- See also: Pirmin Schmid — http://www.pirmin-schmid.ch